CLINICAL TRIAL: NCT05659290
Title: Alternating Treatment With Fruquintinib and Bevacizumab Plus Capecitabine Versus Bevacizumab Plus Capecitabine as Maintenance Therapy Following First-line Treatment for Metastatic Colorectal Cancer: A Multi-center, Parallel-group, Phase II Study.
Brief Title: Alternating Treatment With Fruquintinib and Bevacizumab Plus Capecitabine as Maintenance Therapy After First-Line Treatment in Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2022-479
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer; Fruquintinib; Bevacizumab; Capecitabine; first-line treatment; Maintenance treatment
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Efficacy of Fruquintinib alternating Bevacizumab plus Capecitabine as maintenance therapy after first-line treatment
  Interventions: Drug: Fruquintinib alternating with Bevacizumab plus Capecitabine
- Arm B (Active Comparator): Efficacy of Bevacizumab plus Capecitabine as maintenance therapy after first-line treatment
  Interventions: Drug: Bevacizumab plus Capecitabine

INTERVENTIONS:
Drug: Fruquintinib alternating with Bevacizumab plus Capecitabine — Maintenance therapy with Fruquintinib 5mg, orally, once daily, d1-14, 2 weeks on/ 1 week off, q3w, followed by Bevacizumab 7.5 mg/kg, iv.gtt,d1,q3w + Capecitabine 850 mg/m2, orally, twice daily, d1-14, q3w; every 6 weeks as a treatment cycle; until unacceptable toxicity, withdrawal of informed consent, death, or other criteria for ending the study (whichever occurs earlier).
  Arms: Arm A
Drug: Bevacizumab plus Capecitabine — Maintenance therapy with Bevacizumab 7.5 mg/kg, iv.gtt,d1,q3w + Capecitabine 850 mg/m2, orally, twice daily, d1-14, q3w; every 3 weeks as a treatment cycle; until unacceptable toxicity, withdrawal of informed consent, death, or other criteria for ending the study (whichever occurs earlier).
  Arms: Arm B

SUMMARY:
This is an open-label, multicenter, randomized parallel-group phase 2 study evaluating the efficacy and safety of Fruquintinib alternating with Bevacizumab plus Capecitabine versus Bevacizumab plus Capecitabine as maintenance therapy following first-line treatment for metastatic colorectal cancer. Approximately 40 patients with metastatic colorectal cancer who have achieved partial remission after completing 8 cycles of standard first-line chemotherapy (FOLFOX combined with Bevacizumab) but are still in un-resectable state will be assigned to 2 maintenance treatment groups by randomization in a 1:1 ratio to receive Fruquintinib alternating with Bevacizumab plus Capecitabine (Arm A) or Bevacizumab plus Capecitabine (Arm B). The study contains a safety lead-in phase in which the safety and efficacy of Fruquintinib alternating with Bevacizumab plus Capecitabine will be assessed in approximately 20 patients. All patients from Arm A and Arm B will be treated until unacceptable toxicity, withdrawal of informed consent, death, or other criteria for ending the study (whichever occurs earlier). The study will evaluate PFS, ORR, DCR, OS and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participated in the study, signed the informed consent, and had good compliance;
2. Age 18-75 (including 18 and 75), gender is not limited;
3. Histologically and/or cytologically confirmed metastatic colorectal cancer (stage IV);
4. The patient with at least one measurable lesion (RECIST 1.1) achieved partial remission after 8 cycles of first-line standard chemotherapy (FOLFOX combined with bevacizumab), and the disease remained in an unresectable state.
5. ECOG performance status of 0-2 points;
6. Expected survival ≥12 weeks;
7. Blood test (without blood transfusion within 14 days) 1) Neutrophil absolute value ≥1.5×10^9/L, platelet ≥100×10^9/L, hemoglobin ≥90g/L); 2) Liver function test (aspartate aminotransferase and glutamate aminotransferase ≤3×ULN, bilirubin ≤1.5×ULN; In case of liver metastasis, AST and ALT≤5×ULN); 3) Renal function (serum creatinine ≤1.5×ULN, or creatinine clearance (CCr)≥60ml/min);
8. Men and women of childbearing age must use effective contraceptive methods.

Exclusion Criteria:

1. Received major surgery within 4 weeks prior to the first drug administration; radiotherapy, radiofrequency ablation, chemotherapy, immunotherapy or molecular targeted therapy for tumors within 2 weeks, and other investigational drugs;
2. Previously received anti-vascular small-molecule targeted drug therapy, such as fuquinitinib, regofenib, etc.;
3. A history of severe intolerance to bevacizumab and capecitabine or 5-Fu (i.e., grade 4 toxicity of one of these drugs; Class 3-4 toxicity of other co-administered drugs is not excluded);
4. Known brain or meningeal metastases:
5. Have hypertension that is not well controlled by antihypertensive medications (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);
6. Obvious clinical bleeding symptoms or obvious bleeding tendency and hemoptysis within 3 months prior to treatment. Or treatment of venous/venous thrombosis events within the preceding 6 months, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism; Long-term anticoagulant therapy with warfarin or heparin, or long-term antiplatelet therapy (aspirin ≥300 mg/day or clopidogrel ≥75 mg/day) is required;
7. Active heart disease, including myocardial infarction, severe/unstable angina in the 6 months prior to treatment. Echocardiography showed that the left ventricular ejection fraction was less than 50%, indicating poor arrhythmia control.
8. The patient had other malignancies (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix) within the previous 5 years or at the same time;
9. Known allergy to the study drug or any of its excipients;
10. Severe active infection or uncontrolled infection;
11. Any other disease, a clinically significant metabolic abnormality, abnormal physical examination or abnormal laboratory examination, for which, in the investigator's judgment, there is reason to suspect that the patient has a disease or condition unsuitable for the use of the investigational agent;
12. Urine routine indicated urine protein ≥2+, and 24 hours urine protein quantity >1.0g.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | 3 years
  Defined as the time between the onset of PD or death when a patient first receives the study drug, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 3 years
  Defined as the proportion of patients who achieved complete response (CR) or partial response (PR)
Disease Control Rate (DCR) | 3 years
  Defined as the proportion of patients achieving CR, PR, or stable disease (SD).
Overall Survival (OS) | 3 years
  Defined as the time between the patient's first receipt of the study drug to death.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No